CLINICAL TRIAL: NCT00498407
Title: A Phase II Study of CP-4055 as Second Line Therapy in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Jean-Michel Gaullier, Clavis Pharma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-202; Grantor: CDER; IND/IDE Number: NA
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Colorectal Cancer; Colorectal Cancer
Keywords: CP-4055; ELACYT(TM); Cancer; Colorectal cancer; CRC; Second line therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CP-4055 — CP-4055 5 mg/mL for infusion, dose: 200 mg/m2/day, schedule: d1-5 q4, 30 minutes IV infusion
  Other Names: ELACYT (TM)

SUMMARY:
Patients with histologically or cytologically confirmed metastatic colorectal cancer (CRC) who have failed a first-line chemotherapeutic regimen containing oxaliplatin and 5-fluorouracil (5-FU) with or without bevacizumab, with or without other Investigational Medicinal Products (IMPs), will receive CP-4055 200 mg/m2/day intravenously (IV) on Day 1-5 every four weeks until complete response or disease worsening/progressing.

DETAILED DESCRIPTION:
This is a multicentre clinical study conducted in the United Kingdom. It is an open label study designed to investigate objective response rate (RR), the time to progression (TTP) and the duration of tumor response in patients with colorectal cancer when treated with CP-4055. The quantitative and qualitative toxicities of the treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed metastatic CRC who have failed a first-line chemotherapeutic regimen containing oxaliplatin and 5-fluorouracil (5-FU) with or without bevacizumab, with or without other Investigational Medicinal Products (IMPs)
2. Measurable disease according to Response Criteria In Solid Tumours (RECIST)
3. Performance Status 0 - 2 according to ECOG (Eastern Cooperative Oncology Group) Performance Status
4. Age 18 years or more
5. Life expectancy > 3 months
6. Signed informed consent (IC)
7. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to CP-4055 treatment. Nursing patients are excluded.
8. Male and female patients must use acceptable contraceptive methods for the duration of time on study, and males also for 3 months after the last CP-4055 dose
9. Adequate haematological and biological functions

Exclusion Criteria:

1. Known brain metastases
2. Radiotherapy to more than 30 % of bone marrow
3. Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
4. Concomitant treatment with a non-permitted medication:

   * Alternative drugs
   * High doses of vitamins
5. History of allergic reactions to ara-C or egg
6. Any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled inter-current illness including ongoing or active infection)
7. Any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
8. Pregnancy, breastfeeding or absence of adequate contraception for both male and female fertile patients
9. Known positive status for HIV and/or hepatitis B or C
10. Drug and/or alcohol abuse
11. Any reason why, in the investigator's opinion, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
• Objective response rate (RR) | October 2008

SECONDARY OUTCOMES:
• Time to progression (TTP) | October 2008
• Duration of tumor response | October 2008
• Characterize the quantitative and the qualitative toxicities of the CP-4055 treatment in this patient population | October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cassidy, MBChB, MD, Principal Investigator — The Beatson West of Scotland Cancer Centre
Locations (4):
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Foresterhill,, Aberdeen
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Medical Oncology Dept. of Cancer Studies and Molecular Medicine, Leicester Royal Infirmary, Leicester
  - Macmillan Lead Clinician in Gastro-intestinal Cancer Mount Vernon Cancer Centre, Northwood